CLINICAL TRIAL: NCT03973957
Title: Talc Outpatient Pleurodesis With Indwelling Catheter: A Randomized Controlled Trial
Brief Title: Talc Outpatient Pleurodesis With Indwelling Catheter
Acronym: TOPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Wissam Abouzgheib, Physician, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-020
Record Dates: First submitted 2019-05-27; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Pleural Effusion; Pleural Diseases; Malignant Pleural Effusion
Keywords: Pleural effusion; Pleural diseases; Pleurodesis; Malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion; Pleural Diseases; Pleural Effusion, Malignant | interventions — Chest Tubes; Fentanyl; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized and controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm (Active Comparator): If undergoing talc slurry in the control arm, the patient will undergo IPC placement in the pulmonary procedure unit on day one of admission. The IPC will then be connected to a pleur-evac as standard of care protocol for chest tube drainage. At 1-2 hours post-IPC placement a chest x-ray will be obtained to assess for full lung re-expansion. If the lung does not fully expand the patient will be excluded from the study. Once full lung re-expansion has occurred, talc slurry will be ordered and the patient will be given 25 mcg of IV fentanyl. Talc slurry (5 g sterile talc, brand name Steritalc, mixed with 50 cc or sterile normal saline in a syringe, per Cooper University Pharmacy protocol) will be administered via the IPC. The patient will remain in the hospital, with continuous drainage measured daily for 2-5 days, depending on drainage of the effusion.
  Interventions: Device: Indwelling pleural catheter placement; Drug: Fentanyl Citrate; Drug: Talc Slurry
- Intervention Arm (Active Comparator): An indwelling pleural catheter (IPC) will be placed during this visit. After complete drainage of the effusion, a chest x-ray will be done to determine if full lung reexpansion occurs. If there is lack of full lung re-expansion the patient will be excluded from the study at this time. If full lung re-expansion is present, the patient will receive an intravenous line (IV) by our nursing staff for analgesia prior to talc administration and will be pre-treated with 25 mcg of IV fentanyl.
  Talc slurry (5 g sterile talc, brand name Steritalc, mixed with 50 cc or sterile normal saline in a syringe, per Cooper University Pharmacy protocol) will then be administered through the IPC. The IPC will then be connected to a circuit that will consist of the IPC connected to a 4-liter fluid drainage collection bag via a one-way Heimlich valve (picture of set up included in additional documents).
  Interventions: Device: Indwelling pleural catheter placement; Drug: Fentanyl Citrate; Drug: Talc Slurry; Device: Drainage collection bag

INTERVENTIONS:
Device: Indwelling pleural catheter placement — Indwelling pleural catheter placement by interventional pulmonologist
  Other Names: IPC; Pleural catheter; Chest tube
Drug: Fentanyl Citrate — Administration of intravenous fentanyl prior to talc slurry instillation in order to avoid pain associated with talc slurry application
  Other Names: "Pain medication"
Drug: Talc Slurry — Administration of 5 grams of medical grade sterile talc mixed in 50 milliliters of normal saline solution via indwelling pleural catheter for purposes of talc slurry pleurodesis
Device: Drainage collection bag — Attachment of one-way Heimlich valve with drainage collection bag circuit to indwelling pleural catheter after talc slurry application for purposes of drainage and pleurodesis in the outpatient setting rather than the inpatient setting.
  Other Names: "Leg bag"
  Arms: Intervention Arm

SUMMARY:
This study will be a prospective, randomized trial comparing a new protocol to the standard of care. The investigators protocol and the standard of care involves a previously established procedure that will be completed in the investigators pulmonary procedure unit. The study will include using previously, well-established procedures (indwelling pleural catheter placement, talc slurry administration through an indwelling pleural catheter, pleuroscopy with talc poudrage administration) in addition to a new protocol (at home continuous drainage via indwelling pleural catheter).

DETAILED DESCRIPTION:
The study design is a prospective, randomized and controlled trial comparing a new protocol to the standard of care. To the investigators knowledge, there is no similar protocol and this will be a single center, pilot study. The control arm will consist of subjects who meet the inclusion criteria for the study and will receive current standard of care management for paramalignant pleural effusion. This will consist of either an indwelling pleural catheter (IPC) placement with subsequent talc slurry administration and hospital admission for continuous drainage, or schedule medical pleuroscopy with talc insufflation poudrage and subsequent IPC placement for continuous drainage while in the hospital. The intervention arm will consist of subjects who meet the inclusion criteria and then will be scheduled for IPC placement in the pulmonary procedure unit as either an outpatient visit or during their hospital admission (if the subject is already admitted to the hospital and recruited via our inpatient consult service). The subjects in this arm will then go home or back to their original admission status with a drainage bag for continuous drainage on the same day as the procedure. This protocol will utilize a circuit with an IPC connected to a continuous drainage bag via a one-way Heimlich valve. It is important to note that while utilizing this circuit is a new protocol for patients with paramalignant pleural effusions, the protocol is the current standard of care practice for patients with pneumothorax and persistent air leak, and is being utilized regularly for these patients by the investigator's department as standard of care for patient needing long-term chest tubes while at home.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Diagnosis of a paramalignant pleural effusion (defined as a recurrent pleural effusion directly caused by malignancy with known thoracic involvement)
* Estimated life expectancy greater than 3 months
* Full lung re-expansion on chest x-ray after thoracentesis

Exclusion Criteria:

* Age less than 18 years old
* Pregnant or lactating subject
* Any history of prior pleural talc administration
* History of an indwelling pleural catheter placed on the side of the active paramalignant pleural effusion
* Estimated life expectancy less than 3 months
* Active clinical heart failure
* Inability to return for frequent follow up appointments
* Current incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to pleurodesis | Up to one month from placement of indwelling pleural catheter
  Will measure the time to pleurodesis in the individual arms

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Abouzgheib, Principal Investigator — Cooper health system
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No